CLINICAL TRIAL: NCT00494598
Title: The Pharmacokinetics of Opioids and Sedative/Hypnotics During Selective Cerebral Perfusion
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Ervant V. Nishanian, Asst Professor of Clinical, Department of Anethesiology Clinical Operations, Columbia University
Other Study IDs: AAAC2983
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2008-10

CONDITIONS: Aortic Aneurysm
Keywords: opioids, cerebral perfusion, arterial pharmacokinetics
MeSH Terms: conditions — Aortic Aneurysm | interventions — Sufentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sufentanil — 200 mcg intra-arterial one time bolus
  Other Names: sufenta

SUMMARY:
There is a need to understand how long anesthetic drugs last in the brain during surgery on the ascending aorta or aortic arch. Drugs can have a prolonged effect when blood temperature is made cold therefore the influence of temperature needs to be studied. This type of surgery allows us to answer questions about how anesthetic drugs behave when they are given during a routine portion of surgery. Patients will be provided with anesthetic drugs during surgery while on a heart lung machine. After the drug is injected into the heart lung machine it will be delivered to the brain to provide more sleep and pain relief. Immediately after the injection of anesthetic drugs, blood samples will be taken from an existing intravenous line in the neck and plasma drug concentrations measured. This will help us to understand how long drugs last in the brain during this type of surgery.

DETAILED DESCRIPTION:
The purpose of this study is to understand the disposition of sufentanil, midazolam and morphine when the drugs are introduced into the arterial circulation of the brain. Patients undergoing surgery on the ascending aorta or aortic arch often require cessation of blood flow to the organs of the body, while maintaining some degree of blood flow to the brain. In order to achieve organ protection during the circulatory arrest phase of surgery, the body is cooled to a core temperature of 28°C. Various techniques including deep hypothermic circulatory arrest, retrograde cerebral perfusion through the superior vena cava, and partial or bilateral antegrade selective cerebral perfusion have been proposed as means to protect the brain from ischemic injury during surgery on the aortic arch. At our institution selective cerebral perfusion has found success for major aortic surgery. This technique was devised and first employed by DeBakey and associates, to protect the brain during aortic arch surgery with bilateral carotid perfusion [1]. Selective cerebral perfusion requires the surgical construction and placement of a Dacron graft onto the right axillary artery that when connected to a cardiopulmonary bypass machine it will provide 10 ml/kg/min antegrade flow for brain perfusion [2]. Cerebral cooling will also decrease the oxygen demand of the brain. In such a way brain ischemia may be minimized. The nature of major aortic arch surgery requires independent cerebral circulation or selective cerebral perfusion for a finite period of time. The cardiopulmonary bypass machine is allowed to perfuse the brain indirectly by serial flow through the right axillary artery to the innominate artery and finally to the right carotid artery. Any anesthetic drug that is introduced into the cardiopulmonary bypass circuit will be delivered the same way. We will take advantage of this independent circuit to safely deliver anesthetic drugs to the brain via the right carotid artery during surgery.

A prior study that enrolled 6 patients has shown that the anesthetic administration is safe and feasible. Patients had no problems related to anesthesia or surgery. All patients left the hospital in stable condition.

ELIGIBILITY:
Inclusion Criteria:

* The study population will comprise individuals who have elected to undergo aortic arch surgery or re-operative cardiac surgery requiring selective cerebral perfusion.
* Patients will be treated according to the standard medical practice of Columbia University Medical Center.
* Patients will be within 21 to 90 years of age.

Exclusion Criteria:

* Patients having known hypersensitivity to the anesthetic agents being studied will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing aortic arch surgery
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of intra-carotid opioids and sedatives during selective cerebral perfusion | one week

CONTACTS AND LOCATIONS:
Overall Officials: Ervant Nishanian, PhD MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States